CLINICAL TRIAL: NCT01749280
Title: Efficacy of Magnetic Resonance Imaging Using Ultrasmall Superparamagnetic Particles of Iron Oxide to Predict Clinical Outcome in Patients Under Surveillance for Abdominal Aortic Aneurysms
Brief Title: Magnetic Resonance Imaging To Predict Outcomes In Aortic Aneurysms
Status: Terminated | Type: Observational
Why Stopped: Study being continued as a multi centre MA3RS study.The patients will be followed up under MA3RS and AAA PET.
Sponsor: University of Edinburgh (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/R1CARl05; 10336 (Registry Identifier: UKRCN)
Record Dates: First submitted 2012-11-30; First posted 2012-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; MRI; USPIO
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abdominal Aortic Aneurysms: Patients will be recruited from the outpatient AAA surveillance population at the vascular unit in the Royal Infirmary of Edinburgh.Potential participation in the study will be completely asymptomatic from their AAA.

SUMMARY:
The aorta is the main blood vessel that comes out of the heart and distributes blood to the whole body. In some people, the aorta becomes swollen (aneurysm) and bursts, especially as it passes through the abdomen. These 'abdominal aortic aneurysms' often occur without symptoms and can burst or rupture without warning. This usually leads to death and represents the thirteenth commonest cause of death in the United Kingdom. In this study, we are looking at a new technique that can look at the aortic aneurysm using magnetic resonance imaging; a technique that does not require x-rays or radiation. We have recently shown that, using magnetic resonance combined with a new imaging agent USPIO, we can detect 'hotspots' of activity in these aneurysms that seem to predict which aneurysms grow rapidly, and are therefore potentially at risk of rupture. We here propose to conduct a study in Edinburgh that will invite all patients who are under surveillance because of an aneurysm. We will image these patients using this novel technique and see if we can identify which patients burst their aneurysm, have an aneurysm that grows so large it needs to have surgery, or die. This will be important to establish as it will potentially lead to a new way of managing people that could ultimately save lives. This is particularly timely as national screening and surveillance programmes are currently being launched.

DETAILED DESCRIPTION:
HYPOTHESIS We hypothesise that uptake of ultrasmall supraparamagnetic particles of iron oxide into the aortic wall will predict abdominal aortic aneurysm growth and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients with an abdominal aortic aneurysm >40 mm

Exclusion Criteria:

1. Any medical history or clinically relevant abnormality identified on the screening medical examination, vital sign measurement, or clinical laboratory examination that is deemed by the principal investigator and/or designee to make the subject ineligible for inclusion.
2. Subjects with planned AAA surgery.
3. Renal impairment with eGFR of <30 mls/min at screening, history of kidney transplant or history of contrast nephropathy.
4. Women of child-bearing potential without contraception,
5. Collagen-vascular disease.
6. Inability to undergo magnetic resonance or computed tomography scanning,
7. Contraindication to MRI scanning (as assessed by local MRI safety questionnaire) which includes but not limited to:

   * Intracranial aneurysm clips (except Sugita) or other metallic objects,
   * History of intra- orbital metal fragments that have not been removed,
   * Pacemakers, implantable cardiac defibrillators and non-MR compatible heart valves,
   * Inner ear implants,
   * History of claustrophobia in MR.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit 237 patients with abdominal aortic aneurysms from the clinical surveillance programme at the Royal Infirmary, Edinburgh. Inclusion criteria will be patients with an abdominal aortic aneurysm >40 mm on ultrasound scanning. Exclusion criteria will include patients with anticipated or planned abdominal aortic aneurysm repair, women of child-bearing potential without contraception, inability to undergo magnetic resonance or computed tomography scanning, life expectancy of <2 years, and those with any form of collagen-vascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine if uptake ultrasmall superparamagnetic particles of iron oxide as determined by percentage R2* change between pre-and post-constant scan will predict abdominal aortic aneurysm growth and rupture in patients with abdominal aortic aneurysms. | 2 yrs
  The change of R2* signal which is determined by the USPIO uptake within the issues will be used to assess the change between pre-and post contrast MRI scans. The investigators will assess if macrophage activity as determined by USPIO change predicts AAA growth and rupture
Does USPIO uptake as determined by percentage change between pre-and post contrast scan co-relates with FDG PET standardised uptake values or tissue to background ratios. | 2 yrs
  As per ethical approval, we have recruited patients under AAA PET study to look at USPIO correlation with 18F-FDG PET. The cellular inflammation can be assessed by USPIO uptake, whilst the metabolic activity can be determined by 18F-FDG PET. In this study, the investigators will determine if there is a correlation between the these two imaging modalties by comparing the R2* change using MRI and standardised uptake values using FDG PET.

CONTACTS AND LOCATIONS:
Overall Officials: David Newby, MD PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Research Imaging Centre/ NHS LOTHIAN, Edinburgh, United Kingdom